CLINICAL TRIAL: NCT06489418
Title: A Prospective, Control-arm, Site Randomized, Evaluator-blinded, Single-centre, Safety, and Efficacy Study of Test Product "Dew Restore Barrier Repair Cream" in Healthy Adult Human Subjects With Dry and Sensitive Skin.
Brief Title: A Clinical Study to Assess the Safety and Effectiveness of Test Product in Healthy Adult Human Subjects With Dry and Sensitive Skin.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Kayura Effects LLP (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: NB240032-KE
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Dry Skin; Sensitive Skin

STUDY DESIGN:
Intervention Model Description: A prospective, control-arm, site randomized, evaluator-blinded, single-centre, safety, and efficacy study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry and Sensitive Skin (Experimental): Wash the face with the gentle cleanser to remove dirt, and oil and pat dry with the towel| tissue paper. Afterwards take the pea side amount of the test product you finger tips, apply it over the face by small dotes and massage it in circular motion until it absorbed.
  Interventions: Other: Dew Restore Barrier Repair Cream
- Control (No Intervention): Wash the application site with warm water and pat dry with towel| tissue paper.

INTERVENTIONS:
Other: Dew Restore Barrier Repair Cream — Wash the face with the gentle cleanser to remove dirt, and oil and pat dry with the towel| tissue paper. Afterwards take the pea side amount of the test product you finger tips, apply it over the face by small dotes and massage it in circular motion until it absorbed.
  Frequency: Twice a Day Route of Administration: Topical
  Arms: Dry and Sensitive Skin

SUMMARY:
A prospective, control-arm, site randomized, evaluator-blinded, single-centre, safety, and efficacy study of Test Product "Dew Restore Barrier Repair Cream" in healthy adult human subjects with dry and sensitive skin.

DETAILED DESCRIPTION:
A total of 27 Subjects will be enrolled to complete 25 Subjects the study. The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be called telephonically by the recruiting department prior to the enrolment visit. Subjects will be told during screening (prior to enrolment) not to wear any facial make-up on the study visit day. The adult female subjects will be instructed to visit the facility as per the below visits.

* Visit 01 (Day 01): Screening, Enrolment, Baseline Evaluation, On Site Product Usage, Post Usage Evaluation
* Visit 02 (Day 02): Evaluations, Product usage period
* Visit 03 (Day 15 +2 Days): Product Usage Period, Evaluations
* Visit 04 (Day 30 +2 Days): Evaluations, End of Study

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 55 years (both inclusive) at the time of consent.
* Sex: Healthy male and non-pregnant/non-lactating females (Preferably equal).
* Females of childbearing potential must have a self-reported negative pregnancy test.
* Subject are generally in good health.
* Subject with dry and sensitive skin at a time of screening. (Dermatological Assessment)
* Subjects forearm must be free of cuts, tattoos, scratches, abrasions, scars, uneven skin tone, sunburn, excessive tan, excessive hair or open wounds on or near the test sites
* Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
* If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
* Subjects are willing to give written informed consent and are willing to come for regular follow up.
* Subjects who commit not to use medicated skincare products other than the test product for the entire duration of the study.
* Subject who have not participated in a similar investigation in the past three months.
* Willing to use test product throughout the study period.

Exclusion Criteria:

* History of any dermatological condition of the skin diseases.
* Subject with present condition of allergic response to any cosmetic product.
* Subject having allergic response to the ink.
* Subjects under chronic medication (e.g. aspirin-based products, anti-inflammatories, anti-histamines, corticotherapy etc.) that might influence the outcome of the study.
* Subject having acne of severe incidence (presence of nodules, cysts or numerous pustules) which requires pharmaceutical or cosmeceuticals, herbal treatment.
* Subjects who have applied topical treatment for at least 4 weeks and any systemic treatment for at least 3 months, before they participated in the study.
* History of alcohol or drug addiction.
* Subjects using other marketed products during the study period.
* Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.
* Pregnant or breastfeeding or planning to become pregnant during the study period.
* History of chronic illness which may influence the cutaneous state.
* Subjects participating in other similar cosmetics, devices or therapeutic trials or skincare products within the last four weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Change in DASI Score (Dry Skin/ichthyosis area and severity index). In scoring scale 0 indicates none and 4 indicates extreme. | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days).
  1. To evaluate the effectiveness of the test product in terms of change in DASI score from the baseline before and after usage of the test product.
Change in Dry Skin Score. In scoring scale 0 indicates absent and 4 indicates Dominated by large scales, advanced roughness, redness present, eczematous changes and cracks. | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days).
  2. To evaluate the effectiveness of the test product in terms of change in overall dry skin score (ODS) from the baseline before and after usage of the test product.
Change in PGA Score. In scoring scale 0 means No appearance and 7-9 means severe. | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days).
  3. To evaluate the effectiveness of the test product in terms of change in PGA score from the baseline before and after usage of the test product.
Change in Skin Hydration | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days).
  4. To evaluate the effectiveness of the test product t in terms of change in skin hydration from the baseline before and after usage of the test product.
Change in Skin Barrier Function | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days).
  5. To evaluate the effectiveness of the test product in terms of change in skin barrier function from the baseline before and after usage of the test product.
Change in skin roughness | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days).
  6. To evaluate the effectiveness of the test product in terms of change in skin roughness from the baseline before and after usage of the test product.
Change in skin scaliness | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days).
  To evaluate the effectiveness of the test product in terms of change in skin scaliness from the baseline before and after usage of the test product.
Change in skin smoothness | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days).
  To evaluate the effectiveness of the test product in terms of change in skin smoothness from the baseline before and after usage of the test product.
Change in skin wrinkles | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days).
  To evaluate the effectiveness of the test product in terms of change in skin wrinkles from the baseline before and after usage of the test product.

SECONDARY OUTCOMES:
Change in desquamation index | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days)
  1. To assess the effectiveness of the test product in terms of change in desquamation index from baseline before and after usage of the test product.
Change in visual assessment of skin dryness. 0 means absent and 4 means very severe | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days)
  2. To assess the effectiveness of the test product in terms of change in visual assessment of skin dryness from the baseline before and after usage of the test product.
Change in Product Perception Questionnaire. 0 means absent and 4 means very severe | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days)
  3. To assess the effectiveness of the test product in terms of subject perception questionnaire after usage of the test product from baseline before and after usage of the test product.
Change in visual assessment of skin smoothness. 0 means absent and 4 means very severe | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days)
  To assess the effectiveness of the test product in terms of change in visual assessment of skin smoothness from the baseline before and after usage of the test product.
Change in visual assessment of skin roughness. 0 means absent and 4 means very severe | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days)
  To assess the effectiveness of the test product in terms of change in visual assessment of skin roughness from the baseline before and after usage of the test product.
Change in visual assessment of skin redness. 0 means absent and 4 means very severe | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days)
  To assess the effectiveness of the test product in terms of change in visual assessment of skin roughness from the baseline before and after usage of the test product.
Change in visual assessment of skin itchiness. 0 means absent and 4 means very severe | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days)
  To assess the effectiveness of the test product in terms of change in visual assessment of skin itchiness from the baseline before and after usage of the test product.
Change in visual assessment of skin scaliness. 0 means absent and 4 means very severe | on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 02 [post 24 (+2) hours of the application], Day 15 (+2 Days) and Day 30 (+2 Days)
  To assess the effectiveness of the test product in terms of change in visual assessment of skin scaliness from the baseline before and after usage of the test product.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd
Locations (1):
- NovoBliss Research Pvt.Ltd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No